CLINICAL TRIAL: NCT00950924
Title: Use of Multifocal Contact Lenses to Stimulate Axial Elongation in Axial Hyperopia
Brief Title: Optical Defocus to Stimulate Eye Elongation in Hyperopia
Acronym: ODSEEH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aller, Thomas A., OD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCT00950924
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Hyperopia; Refractive Error
Keywords: Hyperopia; Refractive Error; Ocular Biometrics; Axial Length; Contact Lenses; Bifocal Contact Lenses
MeSH Terms: conditions — Hyperopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bifocal Contact Lenses (Experimental): Simultaneous Vision Bifocal Soft Contact Lenses will be prescribed such that the distance vision as measured by manifest subjective refraction will be properly corrected by the near vision add power and undercorrected by the distance power.
  Interventions: Device: Simultaneous Vision Bifocal Soft Contact Lenses
- Single Vision Soft Contact Lenses (Placebo Comparator): Subjects will be fitted with single vision soft contact lenses with goal of corrected emmetropia at a distance of 20 feet.
  Interventions: Device: Single Vision Soft Contact Lenses

INTERVENTIONS:
Device: Simultaneous Vision Bifocal Soft Contact Lenses — Simultaneous Vision Bifocal Soft Contact Lenses will be prescribed such that the distance vision as measured by manifest subjective refraction will be properly corrected by the near vision add power and undercorrected by the distance power.
  Arms: Bifocal Contact Lenses
Device: Single Vision Soft Contact Lenses — Single vision soft contact lenses will be prescribed to properly correct the distance vision as measured by manifest subjective refraction.
  Arms: Single Vision Soft Contact Lenses

SUMMARY:
Axial hyperopia results when the length of the eye is too short for the eye to properly focus distance objects on the retina while the focusing system is relaxed. Emmetropization is the process by which the eye actively adjusts various components of the eye to gradually improve the focus of the eye. Emmetropization frequently involves either an increase or a decrease in the growth of the eye, particularly during infancy and childhood. Numerous animal studies suggest that if an animal is exposed to retinal images located behind the retina either centrally or peripherally, the eye will grow in the direction of the focused image. If an abnormally short eye has resulted in hyperopia, exposing such an eye to retinal images partially located behind the retina might encourage axial elongation, thus reducing the hyperopia.

DETAILED DESCRIPTION:
Hyperopia or farsightedness may cause distance vision and near vision to be blurred. Depending on the severity of the condition and the age of the patient and the status of the binocular vision system, hyperopia can also cause fatigue, asthenopia, headaches, double vision, and amblyopia. Low to moderate amounts of hyperopia rarely cause much difficulty in the young person, but will eventually cause significant near vision problems as the patient ages. Hyperopia can be caused by the eye being too short (axial hyperopia) or by the cornea being too flat or the crystalline lens being to weak (refractive hyperopia). It has been established by the PI that axial growth can be dramatically lessened in children and adolescents with myopia through the use of bifocal contact lenses prescribed in a particular way (The CONTROL Study). Studies by Earl Smith, O.D., Ph.D. have suggested that multi-zonal contact lenses that provide proper axial focus while manipulating peripheral defocus can either discourage or encourage axial growth to treat myopia or hyperopia respectively. In the present study, simultaneous vision bifocal soft contact lenses will be used to encourage axial growth in hyperopic children and adolescents with axial hyperopia in an effort to reduce hyperopia. Subjects will be randomly assigned to wear either bifocal soft contact lenses or single vision soft lenses. The bifocal contact lenses will be prescribed to provide for clear central vision at both distance and near with the near zone of the contact, thus exposing the retina to hyperopic defocus from the distance zone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-12
* Hyperopia > +1.25 each eye (cycloplegic refraction)
* Ability to wear soft contact lenses

Exclusion Criteria:

* Amblyopia
* Strabismus
* Astigmatism > 1.00 diopters
* Axial Length > 24.00 mm

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-10 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Axial length | One year

SECONDARY OUTCOMES:
Refractive Error | One year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Aller, O.D., Principal Investigator — Unafilliated
Locations (1):
- 711 Kains Ave, San Bruno, California, United States